CLINICAL TRIAL: NCT00565591
Title: A Stepwise, Rising Dose Study of Male Subjects With Mild Intermittent Asthma to Assess the Topical Safety and Tolerability of Albuterol Sulfate Acu-30™ DPI Compared With Placebo Acu-30™ DPI
Brief Title: Study Mild Intermittent Asthma to Assess the Topical Safety and Tolerability of Albuterol Sulfate Acu-30™ DPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respirics Inc. (Industry)
Responsible Party: Andre van As MD PhD, Respirics Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RA1101C
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Allergic Asthma
Keywords: asthma; inhaler device; albuterol sulfate
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Placebo Comparator)
  Interventions: Drug: Albuterol sulfate

INTERVENTIONS:
Drug: Albuterol sulfate — Single dose dry powder by inhalation

SUMMARY:
This open label single blind study will determine the safety of albuterol sulfate dry powder in a novel inhaler by observing for the potential occurrence of reflex bronchial constriction after inhalation of increasing doses of the compound.

DETAILED DESCRIPTION:
This is a single blind (investigator unblinded), open label, single exposure, non-randomized, single center, outpatient, stepwise, rising dose study in male subjects with mild intermittent asthma to assess topical safety and tolerability of Albuterol Sulfate Acu-30™ DPI, compared with Placebo Acu-30™ DPI. Increasing doses of each drug will be administered in a sequential fashion in 4 steps to 3 different subjects at each step (a total of 12 subjects) with mild intermittent asthma in each step.

ELIGIBILITY:
Inclusion Criteria

* Mild intermittent asthma (meeting GINA specifications - www.ginasthma.com)
* Medically normal subjects with no significant abnormal findings
* No tobacco (nicotine products) use for at least 2 years before the study starts
* Normal (or abnormal and clinically insignificant) laboratory values at screening (potassium or glucose levels)
* No significant medical or surgical conditions (COPD, cystic fibrosis, severe allergic rhinitis)

Exclusion Criteria:

* Past or present history of experiencing any allergic reaction to the medications/formulations administered in this study, or in the opinion of the Principal Investigator, suggests an increased potential for an adverse hypersensitivity
* Subject with abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Principal Investigator

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of Albuterol Sulfate Acu-30™ DPI compared with Placebo Acu-30™ DPI in male volunteers with mild intermittent asthma. | 3 hours

SECONDARY OUTCOMES:
To perform an exploratory assessment of the pharmacokinetics (PK) of a single dose of Albuterol Sulfate Acu-30™ in a limited population of male volunteers with mild intermittent asthma. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Holly Brown, MD, Principal Investigator — Private practise
Locations (1):
- Iowa Clinical Research Corporation, Iowa City, Iowa, United States